CLINICAL TRIAL: NCT02777476
Title: Clinical Performance of B-Lite® Light Weight Breast Implant
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: G&G Biotechnology Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-010
Record Dates: First submitted 2016-04-21; First posted 2016-05-19 (Estimated); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Breast Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | US Export: No

ARMS (1):
- procedure with B-Lite® Light Weight Breast Implant (Experimental)
  Interventions: Device: B-Lite- Light Weight Breast Implants

INTERVENTIONS:
Device: B-Lite- Light Weight Breast Implants

SUMMARY:
This is a post-marketing study for B-Lite® implants that carry the EC certificate for marketing in Europe and AMAR certificate for marketing in Israel. To date, thousands of implants have already been implanted in women. The study is open for primary augmentation patients only. All surgeries will be performed as per standard practice at the given study site. No parallel surgical procedures will be performed at the same session.

ELIGIBILITY:
Inclusion Criteria:

* Genetic women between the ages of 18 and 60 seeking primary breast augmentation
* Patient is eligible to undergo MRI (i.e., no implanted metal or metal devices, no history of severe claustrophobia)
* Patient provides signed informed consent
* Patient agrees to comply with the study protocol and complete all required follow up visits, including to undergo MRI
* Patient agrees to return the device to the Sponsor should the implant have to be explanted
* The patient has realistic expectations of surgical results after discussion with investigator and is an acceptable candidate for breast augmentation.

Exclusion Criteria:

* Patients with active infection anywhere in their body
* Patient is pregnant or nursing at the time of recruitment, or has been in the 6 months preceding recruitment date, or not willing to use reliable means of contraception during the first year after surgery
* Patient was implanted with any silicone implant other than breast implants (e.g., silicone artificial joints or facial implants)
* Patient breast tissue is clinically incompatible for the procedure (e.g., tissue damage resulting from radiation, insufficient tissue coverage or compromised vascularity)
* Patient has a condition, or is under treatment for any condition, which, in the opinion of the investigator and/or consulting physician(s), may constitute an unwarranted surgical risk (e.g., unstable cardiac or pulmonary problems, possible allergies and/or extraordinary immune response to implant)
* The patient has a history of mental instability and/or history of pharmaceutical psychiatric treatment
* Patient unable to understand the scope of the study and/or surgery
* The patient has any disease, including uncontrolled diabetes (e.g., HbA1c > 8%), that is clinically known to impact wound healing ability
* Patient has existing costal injuries
* Patient has abscesses, malignant tumors (cancer or recurrent metastases), clinically relevant cysts or advanced fibrotic disease or patient with BIRAD ≥3
* Are not willing to undergo further surgery for revision, if medically required
* The patient has a confirmed rheumatic disease or syndrome (e.g., SLE, Sjogren's syndrome, scleroderma, polymyositis or any connective tissue disorder, rheumatoid arthritis, crystalline arthritis, infectious arthritis, spondyloarthropathies, any other inflammatory arthritis, fibromyalgia or chronic fatigue syndrome)
* The patient has a severe breast and upper trunk deformity
* The patient participated in an investigational trial within 90 days of enrollment
* The patient has undergone an invasive medical procedure within 90 days of enrollment.
* Aesthetic addiction, drug abuse, alcohol abuse

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2016-10 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Changes in breast size measurements | 3 years
Changes in bra size measurements | 3 years

CONTACTS AND LOCATIONS:
Locations (3):
- ETHIANUM, Heidelberg, Germany
- Herzelia Medical Center, Herzliya, Israel
- Akademikliniken, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No